CLINICAL TRIAL: NCT05883514
Title: The Feasibility of Motivational Interviewing on Emotional Intelligence, Dispositional Optimism, and Adherence to Care Practices Among Patients With Permanent Pacemaker
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mahmoud Khedr, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0001
Record Dates: First submitted 2023-05-20; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Pacemaker DDD
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Group one (study group, 35 patients): received the Motivational interviewing intervention.
  Interventions: Behavioral: Motivational interviewing
- Control group (No Intervention): Group two(the control group, 35 patients): will receive routine hospital care such as medication administration, assessment of vital signs, and hygienic care.

INTERVENTIONS:
Behavioral: Motivational interviewing — According to the Miller and Rollnick principles, the framework of the motivational interviewing group's sessions was taken from the workbook of the intervention's six sessions of motivational interviewing. A researcher recruited participants in groups of 7 patients for six sessions of 60-90 minutes each (two sessions per week). The training sessions covered topics like stress alleviation, appropriate drug usage, quitting smoking, regular physical activity, healthy eating habits, and regular physical activity. Patients in the control group got standard treatment for PPM, including education on proper medication usage, nutrition, and exercise, as well as regular checking.
  Arms: Intervention group

SUMMARY:
A cardiac pacemaker is an artificial apparatus that stimulates the myocardium electrically to depolarize, to begin a contraction when the heart's natural pacemaker does not work properly. Pacemakers are essential when dysrhythmias or conduction defects compromise the electrical system and the heart's hemodynamic response.

The current status aimed to assess the feasibility of motivational interviewing on emotional intelligence, dispositional optimism, and adherence to care practices among patients with permanent pacemaker.

DETAILED DESCRIPTION:
According to the Miller and Rollnick principles, the framework of the motivational interviewing group's sessions was taken from the workbook of the intervention's six motivational interviewing sessions. A researcher recruited participants in groups of 7 patients for six sessions of 60-90 minutes each (two sessions per week). The training sessions covered stress alleviation, appropriate drug usage, quitting smoking, regular physical activity, healthy eating habits, and regular physical activity. Patients in the control group got standard treatment for PPM, including education on proper medication usage, nutrition, exercise, and regular checking.

ELIGIBILITY:
Inclusion Criteria:

* Patients with permanent cardiac pacemaker implantation aged from 20 up to 65 years old.
* Both sexes (male & female).
* Able to communicate verbally.
* Free from psychotic disorders.
* Not scheduled for other surgeries.
* Agree to participate in the current study.

Exclusion Criteria:

* Patients with severe mental problems

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Adherence with Pacemaker Care Practices | 2 months
  This tool was developed by (Sharma K, 2018) to assess adherence of the patients to pacemaker care practices. It was adapted and translated into Arabic language by the researcher. It included 15 items related to patients' adherence to care practices of pacemaker .
Emotional Intelligence | 2 months
  Emotional Intelligence Scale by (Schutte et al., 1998) to assess the level of emotional intelligence. This scale consists of 33 items, which can be divided into 4 main subscales (perception of emotion, managing own emotions, managing others' emotions, and utilization of emotion).
Dispositional optimism | 2 months
  The original LOT-R is a self-report questionnaire, measuring dispositional optimism and developed by (Scheier, Carver, & Bridges, 1994). The questionnaire consists of 10 items, of which three positively formulated items (1, 4, and 10), three negatively formulated items (3, 7, and 9), and four "filler" items (2, 5, 6, and 8).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khedr MA, Ali EA, Sanhoury MI, Hussein RM. The feasibility of motivational interviewing on adherence to care practices, emotional intelligence, and dispositional optimism among patients with permanent pacemakers. Eur J Cardiovasc Nurs. 2024 Jul 19;23(5):497-509. doi: 10.1093/eurjcn/zvad113. PMID 38165278